CLINICAL TRIAL: NCT01659645
Title: Amino Acid Transport Imaging of Breast Carcinoma Via Anti-3-[18F]FACBC PET-CT: A Pilot Study
Brief Title: Anti-1-amino-3-[18F]Fluorocyclobutyl-1-carboxylic Acid (Anti-[18F](FACBC)Positron Emission Tomography (PET-CT) of the Breast
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, David M. Schuster, MD, Sponsor-Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00052551; FACBCBr (Other: Other)
Record Dates: First submitted 2012-08-01; First posted 2012-08-08 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FACBC (Experimental)
  Interventions: Drug: FACBC

INTERVENTIONS:
Drug: FACBC — Drug FACBC will be given intravenously (IV) over 2 minutes prior to performing the PET scan

SUMMARY:
Breast carcinoma is the most frequent cancer in women, affecting an estimated 207,090 in 2010 leading to 39,840 cancer related deaths.

Fludeoxyglucose F 18 Injection (FDG) Positron Emission Tomography, (PET) or PET-CT has become the a standard method for isolating the tumor. However, FDG is insensitive in small breast tumors and certain histologic types such as lobular, certain types of breast carcinoma. In addition, FDG uptake can be nonspecific since inflammatory some benign lesions may also evidence have accumulation of this radiotracer. Hence there is a need for a tracer/imaging tool that increases the ability to characterize detect breast carcinoma and to detect locoregional spread, as well as monitor therapeutic treatment response.

anti-3-[18F]. anti-1-amino-3-[18F]fluorocyclobutyl-1-carboxylic acid (FACBC) is an amino acid based PET radiotracer which has shown utility in detecting a variety of tumors. In cell culture experiments,FACBC has shown uptake in the breast tumor cell line.

The primary aim of this study is to determine if FACBC PET-CT demonstrates uptake within breast carcinoma (primary site and/or locoregional lymph nodes) and to study uptake kinetics via time-activity curves from dynamic imaging characteristics. The investigators will enroll 12 patients who have a breast mass or masses and/or lymph nodes naïve to therapy about to undergo biopsy or post-biopsy pre-therapy. All patients will undergo standard of care imaging as appropriate such as mammography, ultrasound, MR, and/or FDG PET-CT scanning. The investigators will then compare findings to determine if this radiotracer is worthy of further study in a more comprehensive experiment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Patients will have a breast mass and/or lymph nodes naïve to therapy about to undergo biopsy or post-biopsy pre-therapy. Patients with known or suspected recurrent disease will be eligible for this protocol.
3. Ability to lie still for PET scanning
4. Patients must be able to provide written informed consent

Exclusion Criteria:

1. Age less than 18.
2. Inability to lie still for PET scanning.
3. Cannot provide written informed consent.
4. Current therapy for breast carcinoma.
5. Positive serum or urine pregnancy test within 24 hours of study.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Presence of FACBC radiotracer in breast carcinoma on FACBC PET scan | Outcomes will be assessed at the end of one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States